CLINICAL TRIAL: NCT03950102
Title: Prospective Study of Stereotactic Body Radiation Therapy as a Bridging Therapy for Hepatocellular Carcinoma Patients on Waiting List for Liver Transplantation
Brief Title: SBRT as Bridging Therapy for Hepatocellular Carcinoma Patients on Transplant Waitlist
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Tiffany Cho-Lam Wong, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW15-191
Record Dates: First submitted 2019-05-02; First posted 2019-05-15 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT (Experimental): SBRT will be used as the primary bridging therapy for HCC patients on waitlist
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Radiation dose of 27.5-50Gy in 5 fractions over 5-14 days with a radical dose as high as achievable based on mean liver dose (MLD), while fulfilling the dose constraints of OARs

SUMMARY:
This is a single center, prospective study to assess the efficacy and safety of using stereotactic body radiation therapy (SBRT) as bridging treatment for hepatocellular carcinoma (HCC) patients on transplant waitlist.

DETAILED DESCRIPTION:
The study population includes patients 18 years of age or older with HCC, who are accepted on waiting list for deceased donor liver transplantation (DDLT).

Patient will be assessed in a multidisciplinary committee and they will receive SBRT unless otherwise contraindicated. Patients will undergo SBRT under standard protocol.

Patients with HCC beyond University of California, San Francisco criteria (UCSF) will be removed from waitlist.

ELIGIBILITY:
Inclusion Criteria:

1. Radiological diagnosis of HCC confirmed according to AASLD criteria
2. All patients who are accepted on deceased donor waiting list
3. HCC within UCSF criteria (defined as solitary tumor <=6.5cm OR up to 3 tumors <=4.5cm, total sum <=8cm)

Exclusion Criteria:

1. age <18 year old;
2. Child's C cirrhosis;
3. Eastern Cooperative Oncology Group (ECOG) score >2;
4. presence of extrahepatic metastasis;
5. radiological tumor invasion to portal, hepatic vein or its branches;
6. absolute contraindications to RT (e.g. previous RT to liver);
7. positive pregnancy test;
8. unwilling or unable to adhere to study requirements and procedure;
9. any other condition, in the investigator's judgment, that increases the risk of SBRT or prevents safe trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk of classical radiation induced liver disease (RILD) after SBRT | From time of SBRT to 3 months afterwards
  Defined as elevated liver transaminases >5 times of upper normal limit or worsening of Child's score by >2 within 3 months after SBRT
Rate of transplant complication | From time of transplant to 1 months afterwards
  Perioperative complication will be assessed according to Clavien-Dindo classification

SECONDARY OUTCOMES:
Rate of dropout from transplant waitlist | From time of enrolment to up to 2 years
  All HCC patients on waitlist will be assessed regularly and will be removed from waitlist if HCC stage is beyond UCSF criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Wong, MBChB, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong TC, Lee VH, Law AL, Pang HH, Lam KO, Lau V, Cui TY, Fong AS, Lee SW, Wong EC, Dai JW, Chan AC, Cheung TT, Fung JY, Yeung RM, Luk MY, Leung TW, Lo CM. Prospective Study of Stereotactic Body Radiation Therapy for Hepatocellular Carcinoma on Waitlist for Liver Transplant. Hepatology. 2021 Nov;74(5):2580-2594. doi: 10.1002/hep.31992. Epub 2021 Sep 30. PMID 34091914